CLINICAL TRIAL: NCT01221584
Title: Centralized Pan-Russian Survey on the Undertreatment of Hypercholesterolemia
Acronym: CEPHEUS
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: NIS-CRU-DUM-2010/1
Record Dates: First submitted 2010-10-14; First posted 2010-10-15 (Estimated); Last update posted 2012-03-01 (Estimated); Status verified 2012-02

CONDITIONS: Dyslipidaemia
Keywords: Dyslipidaemia; LDL-C goals; guidelines
MeSH Terms: conditions — Dyslipidemias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Subject 18 years of age or older on lipid lowering drug treatment for at least 3 months, with no dose change for a minimum of 6 weeks..

SUMMARY:
The purpose of the study is to establish the proportion of patients on lipid-lowering pharmacological treatment reaching the LDL-C goals according to the All-Russian Scientific Cardiology Society guidelines/ the 4th Joint European Task Force guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be 18 years of age or older of either gender or race.
* Subject must provide informed consent and comply with the survey procedures.
* Subject is on lipid lowering drug treatment for at least 3 months, with no dose change for a minimum of 6 weeks.

Exclusion Criteria:

* Subjects who are unwilling or unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject on lipid lowering drug treatment for at least 3 months, with no dose change for a minimum of 6 weeks..
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2010-10; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Establish the proportion of patients on lipid-lowering pharmacological treatment reaching the LDL-C goals according to the All-Russian Scientific Cardiology Society guidelines/the Fourth Joint European Task Force guidelines | 1 visit - 1-3 days

SECONDARY OUTCOMES:
Establish the proportion of patients on lipid-lowering treatment reaching the LDL-C goals according to the Russian guidelines in the following sub-populations: Primary/secondary prevention patients, Patients with metabolic syndrome | 1 visit - 1-3 days
Establish the proportion of patients on lipid-lowering treatment reaching the LDL-C goals according to the FJETF/ NCEP ATP III guidelines, in all population and in Primary/secondary prevention patients, Patients with metabolic syndrome | 1 visit - 1-3 days
Establish the proportion of patients on lipid-lowering treatment reaching the non HDL-C goals according to the NCEP ATP III / updated 2004 NCEP ATP III guidelines in the sub-population patients with fasting triglycerides >200 mg/dL (2.26mmol/L) | 1 visit - 1-3 days

CONTACTS AND LOCATIONS:
Overall Officials: Alexey Stepanov, Prof, Study Director — AstraZeneca; Prof. Boytsov, Principal Investigator — RKNPK; Acad Oganov, Principal Investigator — Center of preventive medicine
Locations (8):
- Russia (8):
  - Research Site, Krasnodar
  - Research Site, Moscow
  - Research Site, Nizhny Novgorod
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg
  - Research Site, Samara
  - Research Site, Voronezh
  - Research Site, Yaroslavl